CLINICAL TRIAL: NCT03350425
Title: Duration of Protection From Pneumonia After Pneumococcal Vaccination in Hemodialysis Patients
Acronym: DOPPIO
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Collaborators: German Center for Infection Research (Other)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Prof. Dr., University of Cologne
Other Study IDs: DOPPIO
Record Dates: First submitted 2017-06-06; First posted 2017-11-22 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D; Pneumonia
Keywords: hemodialysis; pneumococcal vaccination
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained for determination of pneumococcal antibody-titers every three months for two years. The samples will be taken on dialysis days and thus constitute only a minimal additional burden for both patients and physicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recently vaccinated patients: Patients who recently received pneumococcal vaccination.
- Patients vaccinated >2 years ago: Patients who received pneumococcal vaccination more than two years ago.

SUMMARY:
The investigators compare two strata of vaccinated patients: those recently vaccinated and those vaccinated more than two years ago. The primary objective is to compare pneumonia rates between the groups. As exploratory objectives, the investigators will describe the anti-pneumococcal antibody titers in hemodialysis patients as a function of time since vaccination, and determine factors influencing antibody kinetics. Further exploratory objectives investigate the relationship between antibody titers and the incidence of pneumonia in hemodialysis patients and extrapolate a possible cut-off for protection from pneumonia.

DETAILED DESCRIPTION:
Participating sites will screen all hemodialysis patients at their outpatient dialysis clinic for eligibility. Eligible patients will be approached and informed by their treating physician. If a patient agrees to participate in the study and to sign an informed consent form, basic data regarding vaccination history, underlying disease, etc. will be entered or electronically imported into the study eCRF. Pneumococcal antibody titers will be drawn at baseline and every 3 months. For newly vaccinated patients baseline titers will be drawn 4 weeks after the vaccination. DZIF CTUs will coordinate titer assessment schedules and inform the participating physicians of upcoming blood samplings. The samples will be taken on dialysis days and thus constitute only a minimal additional burden for both patients and physicians. DZIF CTUs will actively follow up on study patients for 2 years after enrolment. This follow-up will include validation of all hospitalizations and deaths documented in an electronic registry database to assess whether the primary endpoint (pneumonia) occurred. Additionally, dialysis units will be contacted every 6 months to assess if pneumonia occurred, which did not require hospitalization. DZIF CTUs will document titer assessment results in the eCRF. Titers will not be disclosed to the attending physicians because revaccination due to knowledge of titers would produce bias. All therapies and diagnostics including vaccinations will be administered solely as part of clinical routine and as recommended by appropriate guidelines (e.g. RKI STIKO recommendations).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form including enrolment in registry database (QiN-registry)
* Patients with stage 5 chronic kidney disease treated with chronic hemodialysis
* Patients who are either already vaccinated or eligible and willing to be vaccinated against pneumococcal infection in accordance with current STIKO recommendations
* Age of 18 years or older

Exclusion Criteria:

* Patients unwilling/ineligible for vaccination under current STIKO recommendations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult hemodialysis patients vaccinated against pneumococcal infection or eligible and willing to be vaccinated
Sampling Method: Non-Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of pneumonia rates between newly vaccinated hemodialysis patients and those vaccinated against pneumococcal infection more than 2 years ago | 2 years

SECONDARY OUTCOMES:
Pneumococcal antibody kinetics as a function of time since vaccination. | 2 years
  Description of antibody titers in hemodialysis patients as a function of time since vaccination.
Factors influencing antibody kinetics | 2 years
  Determination of factors influencing antibody kinetics (e.g. age, prior or ongoing immunosuppression, medication, prior vaccination history) by multiple multivariate models

OTHER OUTCOMES:
Exploration of the relationship between anti-pneumococcal antibody titers and a possible cut-off for protection from pneumonia | 2 years
  Exploration of the relationship between anti-pneumococcal antibody titers and the incidence of pneumonia in hemodialysis patients and extrapolation of a possible cut-off for protection from pneumonia.
Factors influencing pneumonia and vaccine response | 2 years
  Evaluation of role of patient history (e.g. underlying kidney disease) and clinical course (e.g. prior hospitalizations) on pneumonia and vaccine response.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A Cornely, MD, Principal Investigator — University of Cologne
Locations (12):
- Germany (12):
  - Eberhard Karls University Tübingen, Tübingen, Baden-Wurttemberg
  - Hospital of the Ludwig-Maximilians-University (LMU), Munich, Bavaria
  - The University Hospital Klinikum rechts der Isar - MRI TUM, Munich, Bavaria
  - University Hospital Giessen und Marburg, Giessen site, Giessen, Hesse
  - University Hospital Heidelberg, Heidelberg, Hesse
  - University Hospital Giessen und Marburg, Marburg site, Marburg, Hesse
  - Hannover Medical School, Hanover, Lower Saxony
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - Medical Clinic, Research Center Borstel, Borstel, Schleswig-Holstein
  - University Hospital Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - University Hospital Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mellinghoff S, von Gersdorff G, Bruns C, Albus K, Dimitriou V, Steinbach A, Schaller M, Vehreschild JJ, Cornely OA, Liss BJ. Duration of Protection From Pneumonia After Pneumococcal Vaccination in Hemodialysis Patients (DOPPIO): Protocol for a Prospective Multicenter Study. JMIR Res Protoc. 2023 Jul 12;12:e45712. doi: 10.2196/45712. PMID 37436797